CLINICAL TRIAL: NCT05443620
Title: Effect of Weight Load on Bone Glucose Uptake in Obese Subjects
Brief Title: Weight Load PET (WELPET)
Acronym: WELPET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: WELPET
Record Dates: First submitted 2022-06-29; First posted 2022-07-05 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Wheelchairs

STUDY DESIGN:
Intervention Model Description: All participants will receive both treatments: (1) High load and (2) No load. This at to separate study visits.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High Load (Active Comparator): Participants will be standing with a heavy weight vest (11 percent of body weight).
  Interventions: Device: Weight vest
- No Load (Placebo Comparator): Participants will be sitting.
  Interventions: Device: Wheelchair

INTERVENTIONS:
Device: Weight vest — A vest weighing up to a maximum of 15 kg.
  Arms: High Load
Device: Wheelchair — Wheelchair in which participants will be sitting to reduce loading on lower extremities.
  Arms: No Load

SUMMARY:
Obesity related ailments, such as cardiovascular diseases (CVD) and metabolic disorders are major causes of death in the world. This trial may result in improved understanding of the causes of obesity and obesity-related disorders. Published data show that if a weight is carried by a rodent, this animal will lose body weight and gain an improved glucose control. Recently published data further show comparable results in humans when carrying an additional weight.

The investigators aim to confirm and further investigate these findings in humans. The investigators plan to let obese participants carry weight vests and monitor their change in glucose uptake in different tissues. This to further examine the effects increased axial loading has on glucose metabolism in different parts of the body.

DETAILED DESCRIPTION:
STUDY OBJECTIVES AND ENDPOINTS

Primary objective

1. Determine if standing with a heavy weight vest (high load, i.e. 11 percent of body weight) for 3 hours increase glucose uptake in bone more than sitting (no load) for 3 hours.

   Secondary objectives
2. Determine if standing with a heavy weight vest (high load, i.e. 11 percent of body weight) for 3 hours increase glucose uptake in fat tissue more than sitting (no load) for 3 hours.
3. Determine if standing with a heavy weight vest (high load, i.e. 11 percent of body weight) for 3 hours increase glucose uptake in muscle more than sitting (no load) for 3 hours.

STUDY DESIGN AND PROCEDURES

Overall study design and procedure protocol

This is an interventional, single center, imaging study with a within-subjects design. The aim is to investigate how increased loading affects the glucose uptake in the weight bearing bones measured with whole-body Positron Emission Tomography (PET)/Computed Tomography (CT) imaging together with the Fluorine-18 labeled glucose analog, 2-deoxy-2-[18F]-fluoro-D-glucose (18F-FDG). Glucose uptake in muscle and fat tissues will also be evaluated. All participants will test 2 different conditions with measurements of bone glucose uptake after:

1. No load - Participant in sitting position.
2. High load - Standing with a heavy weight vest consisting of 11 percent of the participants body weight.

Participants will receive loading for 3 hours before measurement with PET/CT imaging. Weight of weight vest are based on participants' body weight at the high load visit. Participants will continue with their normal lifestyle during the whole study. There will be a total of three study visits. Study visits will be on 3 separate days within approximately 3 weeks with a minimum of 2 days between each visit. Visits after screening will occur in a randomised order for all participants. All participants will undergo both study treatments and measurements will be compared within each participant from high load and no load visit.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent to participate in the study.
2. Consent out of free will.
3. 18-65 years of age.
4. Maximum body weight of 115 kg.
5. Obesity as defined by a BMI >30 and ≤35 kg/m2. Fat mass >25 percent of total body weight.
6. Willingness to comply with the study protocol.
7. Confirmation of adequate function of major organs and systems as judged by investigator
8. Normal or clinically non-significant screening of blood samples:

   1. Hemoglobin (Hb), White Blood Cell Count (WBC), thrombocyte count, sodium (Na), potassium (K), chloride (Cl), calcium (Ca), creatinine, aspartate transaminase (AST), alanine transaminase (ALT), alkaline phosphatase (ALP), glycated hemoglobin (HbA1c), fasting blood glucose, C-reactive protein (CRP), free thyroxine (fT4), thyroid stimulating hormone (TSH), Triglycerides, high-density lipoprotein (HDL), low-density lipoprotein (LDL).
   2. Normal or clinically non-significant aberrations of screening blood samples are defined as:

   i. Normal: Values within the reference interval supplied by the Turku University Hospital lab.

ii. Clinically non-significant aberration: as judged by investigator (Clinical significance judged by investigator)

Exclusion Criteria:

1. Chronic disease that could interfere with the participation in the study as judged by the investigator such as neurological, renal, hepatic, endocrine, cardiovascular, pulmonary, hematological, or gastrointestinal disorders.
2. Diagnosed diabetes.
3. Chronic pain such as pain that is constant and impairs quality of life as judged by the investigator; for example: significant back, hip or knee pain.
4. Regular consumption of medications or natural supplements that affect weight, inhibit physical activity or increase the risk of adverse effects as judged by the investigator. The following drugs will not be accepted:

   a. β-blockers, Glucagon-Like Peptide 1 (GLP-1)-agonists, Dipeptidyl Peptidase-IV (DPP-IV)-inhibitors, Sodium-glucose Cotransporter-2 (SGLT2)-inhibitors, sulfonylureas, insulin, orlistat, anti-obesity drugs, antidepressants, bisphosphonates, β2-agonists, intra articular or parenteral corticosteroids, diuretics, benzodiazepines, or central nervous system stimulating drugs such as methylphenidate or dextroamphetamine.
5. Gastric by-pass surgery or equivalent metabolic surgery in the gastrointestinal tract.
6. Reduced mobility as judged by the investigator.
7. Use of any illegal drugs according to local regulations, use of tobacco or nicotine products (e.g. cigarettes or snuff) or consuming excessive amounts of alcohol.

   a. Excessive amounts of alcohol defined as:

   i. Consumption of more than 9 glasses of wine for women, 14 glasses of wine for men (15 cl/glass 11 percent alcohol) or equivalent as judged by the investigator during an ordinary week will not be accepted.
8. Change in body weight of ≥5 kg during the last 3 months.
9. Drastic change in lifestyle during the last 3 months including a significant change in physical activity or dietary habits as judged by the investigator.
10. Apparent risk of not being able to comply with the study protocol for any reason as judged by the investigator.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-11-22 (Actual); Study Completion 2024-11-22 (Actual)

PRIMARY OUTCOMES:
Change in glucose uptake in loaded bones | 3 hours
  Change in ratio between glucose uptake in loaded bones (e.g. femur, tibia) and glucose uptake in not loaded bones (e.g. humerus). Change in ratio (in percent between high load and no load) compared after 3 hours of different interventions.

SECONDARY OUTCOMES:
Change in glucose uptake in loaded fat tissues | 3 hours
  Change in ratio between glucose uptake in loaded fat tissues (e.g. subcutaneous (thigh & abdominal) and visceral) and glucose uptake in not loaded fat tissues (e.g. subcutaneous arm). Change in ratio (in percent between high load and no load) compared after 3 hours of different interventions.
Change in glucose uptake in loaded muscles | 3 hours
  Change in ratio between glucose uptake in loaded muscles (e.g. m. quadriceps femoris, m. hamstrings, m. soleus) and glucose uptake in not loaded muscles (e.g. m. biceps brachii, m. triceps brachii). Change in ratio (in percent between high load and no load) compared after 3 hours of different interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Roivainen, Principal Investigator — Turku University Hospital, Turku PET Centre
Locations (1):
- Turku University Hospital, Turku PET Centre, Turku, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jansson JO, Palsdottir V, Hagg DA, Schele E, Dickson SL, Anesten F, Bake T, Montelius M, Bellman J, Johansson ME, Cone RD, Drucker DJ, Wu J, Aleksic B, Tornqvist AE, Sjogren K, Gustafsson JA, Windahl SH, Ohlsson C. Body weight homeostat that regulates fat mass independently of leptin in rats and mice. Proc Natl Acad Sci U S A. 2018 Jan 9;115(2):427-432. doi: 10.1073/pnas.1715687114. Epub 2017 Dec 26. PMID 29279372
- [Background] Ohlsson C, Gidestrand E, Bellman J, Larsson C, Palsdottir V, Hagg D, Jansson PA, Jansson JO. Increased weight loading reduces body weight and body fat in obese subjects - A proof of concept randomized clinical trial. EClinicalMedicine. 2020 Apr 30;22:100338. doi: 10.1016/j.eclinm.2020.100338. eCollection 2020 May. PMID 32510046
- [Derived] Bellman J, Sjoros T, Hagg D, Atencio Herre E, Hieta J, Eskola O, Laitinen K, Nuutila P, Jansson JO, Jansson PA, Kalliokoski K, Roivainen A, Ohlsson C. Loading Enhances Glucose Uptake in Muscles, Bones, and Bone Marrow of Lower Extremities in Humans. J Clin Endocrinol Metab. 2024 Nov 18;109(12):3126-3136. doi: 10.1210/clinem/dgae344. PMID 38753869